CLINICAL TRIAL: NCT00508937
Title: The Effects of Increased Dietary Protein Intake on Insulin Sensitivity in Stable Weight Individuals, Independent of Dietary Content of Carbohydrate and Saturated Fat
Brief Title: Dietary Protein and Insulin Sensitivity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MM3717
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Insulin Resistance; Type 2 Diabetes; Metabolic Syndrome; Cardiovascular Disease; Dyslipidemia
Keywords: Diet; Protein; Glucose; Insulin; Cholesterol; Triglycerides; LDL subclasses
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Metabolic Syndrome; Cardiovascular Diseases; Dyslipidemias | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator)
  Interventions: Other: Diet
- 2 (Experimental)
  Interventions: Other: Diet
- 3 (Experimental)
  Interventions: Other: Diet
- 4 (Experimental)
  Interventions: Other: Diet
- 5 (Experimental)
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — 15% protein, 55% carbohydrate, 30% fat (7% saturated, 7% polyunsaturated)
  Arms: 1
Other: Diet — 20% protein, 35% carbohydrate, 45% fat (7% saturated, 7% polyunsaturated)
  Arms: 2
Other: Diet — 20% protein, 35% carbohydrate, 45% fat (15% saturated, 7% polyunsaturated)
  Arms: 3
Other: Diet — 30% protein, 35% carbohydrate, 35% fat (7% saturated, 7% polyunsaturated)
  Arms: 4
Other: Diet — 30% protein, 35% carbohydrate, 35% fat (15% saturated, 7% polyunsaturated)
  Arms: 5

SUMMARY:
The overall objective of the Dietary Protein and Insulin Sensitivity Study is to test the hypothesis that increased protein in a diet with reduced carbohydrate (35% energy) can ameliorate insulin resistance in the absence of weight loss, and that this effect is independent of saturated fat content. Moreover, we will test whether such diets result in beneficial changes in total LDL cholesterol, small, dense LDL, and HDL cholesterol that are also independent of saturated fat intake.

DETAILED DESCRIPTION:
Insulin resistance is a major metabolic disturbance associated with excess adiposity that contributes to atherogenic dyslipidemia and predisposes to both cardiovascular disease and type 2 diabetes mellitus. The effects on insulin resistance of changes in dietary macronutrient composition in the absence of weight loss are poorly understood. To better understand these effects, we will study men and women with insulin resistance after 4 weeks on a basal diet (15% protein, 55% carbohydrate, 30% fat) and 4 weeks after random assignment to the basal diet or one of 4 diets with 35% carbohydrate and either 20% or 30% protein, and either 7% or 15% saturated fat. At the end of each dietary period (4 weeks and 8 weeks), we will draw a blood sample for detailed metabolic measurements and measure insulin sensitivity by the frequently sampled intravenous glucose tolerance test (FSIGT) method. In addition to insulin resistance, we will assess the effect of dietary composition on parameters of atherogenic dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 27 and ≤ 40 kg/m2
* HOMA-IR ≥ 2.5
* Non-smoking
* Total cholesterol and LDL cholesterol <95th percentile for sex and age
* Fasting triglycerides < 500mg/dl
* Fasting blood sugar < 126
* Urinary microalbumin < 30 mg/L
* Normal thyroid stimulating hormone levels
* Hematocrit ≥ 36%
* Blood pressure < 150/90
* At least 3 months of a weight-stable state (± 5 lbs) prior to the study. During the study, subjects will be required to maintain their body weight within ± 3% (up to a maximum change of 5 lbs) of their initial weight over the course of any consecutive two weeks after the second week of baseline diet or during the last week of each diet phase

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin cancer) in the last 5 years
* Use of drugs known to affect lipid metabolism or insulin resistance, hormones, or the blood thinning agent, warfarin
* Use of alcohol or dietary supplements during the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity by Frequently Sampled Intravenous Glucose Tolerance test | 4wks and 8wks
Total Cholesterol | 4wks and 8wks
LDL Cholesterol | 4wks and 8wks
HDL Cholesterol | 4wks and 8wks
Triglycerides | 4wks and 8wks
LDL peak particle size | 4wks and 8wks
LDL subclasses | 4wks and 8wks

SECONDARY OUTCOMES:
Apolipoprotein B | 4wks and 8wks
Apolipoprotein A1 | 4wks and 8wks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (2):
- United States (2):
  - Cholesterol Research Center, Berkeley, California
  - San Francisco General Hospital, San Francisco, California

REFERENCES:
- [Derived] Chiu S, Williams PT, Dawson T, Bergman RN, Stefanovski D, Watkins SM, Krauss RM. Diets high in protein or saturated fat do not affect insulin sensitivity or plasma concentrations of lipids and lipoproteins in overweight and obese adults. J Nutr. 2014 Nov;144(11):1753-9. doi: 10.3945/jn.114.197624. Epub 2014 Sep 3. PMID 25332473